CLINICAL TRIAL: NCT00071305
Title: Non-Invasive Seizure Localization in Patients With Medically Refractory Localization Related Epilepsy: Synchronized MEG-EEG Recordings
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040016; 04-N-0016
Record Dates: First submitted 2003-10-17; First posted 2003-10-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-10-06

CONDITIONS: Epilepsy
Keywords: Magnetoencephalography; Electroencephalography; Epilepsy; Dipole Modeling; Surgery
MeSH Terms: conditions — Epilepsy

SUMMARY:
This study will evaluate the magnetoencephalography (MEG) alone and together with electroencephalography (EEG) in non-invasive presurgical evaluation. It will look at the contribution of those methods in determining the location of the epilepsy seizure, compared with doing so through an invasive method. EEG measures electronic potential differences on the scalp. On the other hand, MEG is a non-invasive technique for recording the activity of neurons in the brain, through recording of magnetic fields caused by synchronized neural currents. It has the ability to detect seizures. Because magnetic signals of the brain vary, this technique must balance two key problems: weakness of the signal and strength of the noise. The EEG is sensitive to extra-cellular volume currents, whereas the MEG primarily registers intra-cellular currents. Because electrical fields are quite dependent on the conductive properties of the tissues, and magnetic fields are significantly less distorted by tissue, the MEG has better spatial resolution. There is a great deal of evidence that EEG and MEG provide complementary data about underlying currents of ions.

Patients 18 years of age or older who have epilepsy that is not relieved, and who are considered candidates for surgery and who accept epilepsy surgery, may be eligible for this study.

Before they have surgery, participants will either sit or lie down, with their head in a helmet covering the entire head, with openings for the eyes and ears. Brain magnetic fields will be recorded with a 275-channel OMEGA system. Throughout the session, visual and two-way audio communication will be maintained with the patient. Acquiring data from the participant will be conducted during several sessions, each lasting from 10 to 60 minutes, not exceeding a total of 120 minutes. If the first recording is not of sufficient quality, the patient may have it repeated once or twice.

Those participants who are found to have a clear seizure focus will proceed directly to surgery that is part of their treatment. Those whose seizure focus is ambiguous will proceed to invasive monitoring.

Participants will be followed in the outpatient clinic at intervals of 1, 3, 6, and 12 months. They may periodically undergo reimaging as considered appropriate.

DETAILED DESCRIPTION:
Objective:

We will use magnetoencephalography (MEG) alone, and in combination with EEG (MEG-EEG), to study the contribution of each method and their combination to the localizing yield of the non-invasive pre-surgical evaluation as compared to the invasive method. We will also correlate seizure origin and localizing data with surgical outcome, and, in retrospect, calculate the proportion of patients in whom invasive monitoring could have been avoided.

Study Population:

Participants in this study will be patients with medically refractory localization-related epilepsy who will be undergoing epilepsy surgery as part of their standard clinical care.

Study Design/Methods:

We will use a 275-channel whole-head MEG System (CTF Systems 2001 Inc). Patients will undergo a supine resting MEG-EEG recording prior to any surgical procedure. The resulting data will be integrated with the data obtained during the patient's standard pre-surgical evaluation, and compared with the invasive data obtained during chronic invasive monitoring (if clinically indicated), and/or intra-operative electrocorticography (all patients-standard of care). When analyzing the data, readers will be blinded to the results of the other modality (MEG vs. EEG, non-invasive vs. invasive).

The patients will be followed in the outpatient clinic at 1-, 3-, 6- and 12-month intervals. Surgical outcomes will be graded according to the Engel and International League Against Epilepsy (ILAE) outcome scales.

The findings from this protocol will not in themselves indicate or lead to epilepsy surgery.

Outcomes:

The primary outcome measure will be the proportion of seizure foci detected and delineated both non-invasively and invasively. The secondary outcome measures will be the proportion of patients with seizure foci co-localized invasively and non-invasively, the correlation of the obtained localizing data from both modalities with surgical outcome, and the correlation between the anatomical location of the epileptogenic zone and surgical outcome.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients older than 18 years of age.

Patients of both sexes and any race or ethnicity who have intractable epilepsy who are deemed surgical candidates and accept epilepsy surgery.

EXCLUSION CRITERIA:

Patients younger than 18 years of age.

Pregnant women.

Patients who are not surgical candidates.

Patients who do not accept epilepsy surgery.

Patients with progressive neurological disorders.

Patients who are unable to cooperate adequately with MEG/EEG recordings

Patients who had brain surgery.

Patients unable to understand and sign consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2003-10-17; Primary Completion 2009-10-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Amo C, Saldana C, Hidalgo MG, Maestu F, Fernandez A, Arrazola J, Ortiz T. Magnetoencephalographic localization of peritumoral temporal epileptic focus previous surgical resection. Seizure. 2003 Jan;12(1):19-22. doi: 10.1016/s1059131102001486. PMID 12495644
- [Background] Baumgartner C, Pataraia E, Lindinger G, Deecke L. Neuromagnetic recordings in temporal lobe epilepsy. J Clin Neurophysiol. 2000 Mar;17(2):177-89. doi: 10.1097/00004691-200003000-00007. PMID 10831109
- [Background] Boon P, D'Have M, Vanrumste B, Van Hoey G, Vonck K, Van Walleghem P, Caemaert J, Achten E, De Reuck J. Ictal source localization in presurgical patients with refractory epilepsy. J Clin Neurophysiol. 2002 Oct;19(5):461-8. doi: 10.1097/00004691-200210000-00009. PMID 12477991